CLINICAL TRIAL: NCT02724553
Title: Comparison of Horizontal and Vertical IOL Haptic Orientation in Negative Dysphotopsia.
Brief Title: Comparison of Haptic Orientation in Negative Dysphotopsia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A recent publication answered the study question being asked
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5150345
Record Dates: First submitted 2016-02-26; First posted 2016-03-31 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Negative Dysphotopsia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vertical orientation of Haptic orientation (Other): The orientation of the IOL haptic will be implanted in the vertical position during routine cataract surgery
  Interventions: Device: Acrylic lens implantation
- Horizontal orientation of Haptic orientation (Other): The orientation of the IOL haptic will be implanted in the horizontal position during routine cataract surgery
  Interventions: Device: Acrylic lens implantation

INTERVENTIONS:
Device: Acrylic lens implantation

SUMMARY:
Previous studies attempted to understand the dysphotopsia phenomenon by examining intraocular lens type, anterior capsule depth, iris-to-lens depth, lens refractive material, clear cornea incision wounds and anterior capsulorrhexis. However, there is limited literature in understanding haptic orientation and negative dysphotopsia; postulated theories and anecdotal reports relate to horizontal haptic orientation and the lateralization of rays such that light is received both in smaller width and anterior to the peripheral retina; however, no formal studies currently exist.

ELIGIBILITY:
Inclusion Criteria: Patients with bilateral cataracts that are visually significant meeting standard criteria for removal and select standard monofocal lens implantation.

Exclusion Criteria: Patients with any prior refractive surgery including prior cataract surgery, corneal ocular pathology, iris atrophy/damage, retinal or optic nerve pathology. Patients with history of peripheral vision loss. Patients selecting multifocal or toric lens implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Presence of negative dysphotopsia after cataract surgery at 6 months | 6 months
  Presence of negative dysphotopsia in the vertical IOL placement compared to horizontal IOL placement

SECONDARY OUTCOMES:
Presence of negative dysphotopsia after cataract surgery at 1 week | 1 week
  Presence of negative dysphotopsia in the vertical IOL placement compared to horizontal IOL placement
Presence of negative dysphotopsia after cataract surgery at 1 month | 1 month
  Presence of negative dysphotopsia in the vertical IOL placement compared to horizontal IOL placement

CONTACTS AND LOCATIONS:
Overall Officials: Howard D Guan, MD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holladay JT, Zhao H, Reisin CR. Negative dysphotopsia: the enigmatic penumbra. J Cataract Refract Surg. 2012 Jul;38(7):1251-65. doi: 10.1016/j.jcrs.2012.01.032. PMID 22727295
- [Background] Narvaez J, Banning CS, Stulting RD. Negative dysphotopsia associated with implantation of the Z9000 intraocular lens. J Cataract Refract Surg. 2005 Apr;31(4):846-7. doi: 10.1016/j.jcrs.2004.08.059. PMID 15899465
- [Background] Masket S, Fram NR. Pseudophakic negative dysphotopsia: Surgical management and new theory of etiology. J Cataract Refract Surg. 2011 Jul;37(7):1199-207. doi: 10.1016/j.jcrs.2011.02.022. PMID 21700100
- [Background] Vamosi P, Csakany B, Nemeth J. Intraocular lens exchange in patients with negative dysphotopsia symptoms. J Cataract Refract Surg. 2010 Mar;36(3):418-24. doi: 10.1016/j.jcrs.2009.10.035. PMID 20202539
- [Background] Osher RH. Negative dysphotopsia: long-term study and possible explanation for transient symptoms. J Cataract Refract Surg. 2008 Oct;34(10):1699-707. doi: 10.1016/j.jcrs.2008.06.026. PMID 18812121
- [Background] Burke TR, Benjamin L. Sulcus-fixated intraocular lens implantation for the management of negative dysphotopsia. J Cataract Refract Surg. 2014 Sep;40(9):1469-72. doi: 10.1016/j.jcrs.2013.11.037. Epub 2014 Jun 20. PMID 24957929
- [Background] Trattler WB, Whitsett JC, Simone PA. Negative dysphotopsia after intraocular lens implantation irrespective of design and material. J Cataract Refract Surg. 2005 Apr;31(4):841-5. doi: 10.1016/j.jcrs.2004.12.044. PMID 15899464
- [Background] Cooke DL. Negative dysphotopsia after temporal corneal incisions. J Cataract Refract Surg. 2010 Apr;36(4):671-2. doi: 10.1016/j.jcrs.2010.01.004. PMID 20362862